CLINICAL TRIAL: NCT02898025
Title: Low Level Laser Therapy and Interferential Current in Patients With Knee Osteoarthritis: Randomized Controlled Trial
Brief Title: Low Level Laser Therapy and Interferential Current in Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Cidade de Sao Paulo (Other)
Responsible Party: Principal Investigator, Richard Eloin Liebano, Principal Investigator, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RLiebano
Record Dates: First submitted 2016-04-20; First posted 2016-09-13 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Electric Stimulation Therapy; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- G1 (Active IFC and Active Laser) (Active Comparator): 42 patients with knee (s) osteoarthritis. All patients will receive guidance on the disease and on joint protection and energy conservation over a period of 50 minutes in a single session. This group (G1) will receive the treatment of Active Interferential Current and Active Laser for 12 sessions.
  Interventions: Device: Active Interferential Current; Device: Active Laser
- G2 (Active IFC and Placebo Laser) (Active Comparator): 42 patients with knee (s) osteoarthritis. All patients will receive guidance on the disease and on joint protection and energy conservation over a period of 50 minutes in a single session. This group (G2) will receive the treatment of Active Interferential Current and Placebo Laser for 12 sessions.
  Interventions: Device: Active Interferential Current; Device: Placebo Laser
- G3 (Placebo IFC and Active Laser) (Active Comparator): 42 patients with knee (s) osteoarthritis. All patients will receive guidance on the disease and on joint protection and energy conservation over a period of 50 minutes in a single session. This group (G3) will receive Placebo Interferential Current and Active Laser for 12 sessions.
  Interventions: Device: Active Laser; Device: Placebo Interferential Current
- G4 (Placebo IFC and Placebo Laser) (Placebo Comparator): 42 patients with knee (s) osteoarthritis. All patients will receive guidance on the disease and on joint protection and energy conservation over a period of 50 minutes in a single session. The placebo group (G4) will receive Placebo Interferential Current and Placebo Laser for 12 sessions.
  Interventions: Device: Placebo Interferential Current; Device: Placebo Laser

INTERVENTIONS:
Device: Active Interferential Current — Involves the application of medium frequency alternating currents
  Other Names: interferential therapy; IFC
  Arms: G1 (Active IFC and Active Laser); G2 (Active IFC and Placebo Laser)
Device: Active Laser — Involves the application of low level laser over the knee
  Other Names: low level laser therapy
  Arms: G1 (Active IFC and Active Laser); G3 (Placebo IFC and Active Laser)
Device: Placebo Interferential Current — It is a sham interferential therapy
  Arms: G3 (Placebo IFC and Active Laser); G4 (Placebo IFC and Placebo Laser)
Device: Placebo Laser — It is a sham laser therapy
  Arms: G2 (Active IFC and Placebo Laser); G4 (Placebo IFC and Placebo Laser)

SUMMARY:
This study aims to evaluate the effectiveness of the low level laser therapy and interferential current in 168 patients with knee osteoarthritis

DETAILED DESCRIPTION:
Interventional

ELIGIBILITY:
Inclusion Criteria:

* History of osteoarthritis of the knee characterized by pain of mild or moderate intensity
* Radiographic evidence of grade 2 or 3 osteoarthritis based on the Kellgren and Lawrence radiographic entry criteria
* Patients with knee osteoarthritis (s) according to the ACR criteria
* VAS 3 to 8
* 5 to 12 Lequesne
* No complaint of pain in other joints of the lower limbs
* Without neurological and cognitive disorders
* No loss of sensation in the lower limbs
* No surgery on the knee (s) in the last 6 months
* Pain symptoms for at least 6 months
* No infiltrations (s) knee (s) in the last 4 weeks
* No use of analgesics 4 hours before treatment

Exclusion Criteria:

* Individuals younger than 18 and older than 80 years
* Complaints from other diseases of the lower limbs, knee prosthesis and / or hip joint instabilities and / or surgery in lower limbs, heart disease, uncontrolled hypertension and diabetes, coagulation disorders in anticoagulant therapy, pregnant women, fibromyalgia and individuals who can not perform isokinetic test who have difficulty performing the TUG, and those that are experiencing abnormal sensitivity to algometry

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2015-11; Primary Completion 2017-03 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Pain intensity measured by a numeric pain scale ranging from 0 to 10. | 4 weeks
Pressure Pain Threshold measured by a pressure algometer. Pressure will be recorded in kPa. | 4 weeks

SECONDARY OUTCOMES:
TUG (Timed Up & Go Test) | Measure at baseline, 4 weeks, 3 months, 6 months
Isokinetic Muscle Assessment | Measure at baseline, 4 weeks, 3 months, 6 months
LeQuesne Questionnaire | Measure at baseline, 4 weeks, 3 months, 6 months
WOMAC (Western Ontario and McMaster Universities Arthritis Index) | Measure at baseline, 4 weeks, 3 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Liebano, PhD, Principal Investigator — Universidade Cidade de Sao Paulo
Locations (1):
- UNICID, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alqualo-Costa R, Thome GR, Perracini MR, Liebano RE. Low-level laser therapy and interferential current in patients with knee osteoarthritis: a randomized controlled trial protocol. Pain Manag. 2018 May;8(3):157-166. doi: 10.2217/pmt-2017-0057. Epub 2018 May 3. PMID 29722602